CLINICAL TRIAL: NCT01624129
Title: New Serological Markers for Eosinophilic Esophagitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: 2011_0023
Record Dates: First submitted 2011-02-08; First posted 2012-06-20 (Estimated); Last update posted 2025-01-09 (Actual); Status verified 2013-01

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Fluticasone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- eosinophilic esophagitis: patients with histopathological defined eosinophilic esophagitis
  Interventions: Drug: Fluticasone

INTERVENTIONS:
Drug: Fluticasone — Guideline-based treatment with fluticasone 0,5 ml (1-0-1), step-up or step-down after 3 months based on the histopathological findings

SUMMARY:
The purpose of the study is to investigate if serological parameters such as "extracellular Serum-Tryptase (ST)" and "eosinophilic cationic protein (ECP)" are useful for the diagnosis and surveillance of the eosinophilic esophagitis (EE).

DETAILED DESCRIPTION:
The eosinophilic esophagitis (EE) is chronic inflammatory and immunological disease. The diagnosis of EE is based upon large numbers of eosinophils in the esophagus on histopathologic examination (> 20 eosinophils per high powered field in at least one specimen) despite acid suppression with a Proton-Pump-Inhibitor (PPI) for at least two weeks.

There are no diagnostic serological markers for EE so far, so that the purpose of the study is to investigate serological markers which are established in other allergic diseases.

ELIGIBILITY:
Inclusion Criteria:

* histopathological defined eosinophilic esophagitis
* Age: 18-80

Exclusion Criteria:

* missing consent form
* contraindications for performing esophagogastroscopy/taking biopsies of the esophagus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monther Bajbouj, MD, Principal Investigator — Technical University of Munich, 2nd Medical Department
Locations (1):
- II. Medical Department, Technical University Munich, Munich, Bavaria, Germany

REFERENCES:
- [Derived] Schlag C, Pfefferkorn S, Brockow K, Haller B, Slotta-Huspenia J, Schulz S, von Werder A, Ring J, Schmid RM, Bajbouj M. Serum eosinophil cationic protein is superior to mast cell tryptase as marker for response to topical corticosteroid therapy in eosinophilic esophagitis. J Clin Gastroenterol. 2014 Aug;48(7):600-6. doi: 10.1097/01.mcg.0000436439.67768.8d. PMID 24177377